CLINICAL TRIAL: NCT01508104
Title: A Dose Escalation, Single Arm, Phase 1b-2 Combination Study of BEZ235 With Everolimus to Determine the Safety, Pharmacodynamics and Pharmacokinetics in Subjects With Advanced Solid Malignancies
Brief Title: Safety Study of BEZ235 With Everolimus in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: funding
Sponsor: University of Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, John Morris, Professor, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBEZ235ZUS08T
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Cancer
Keywords: solid tumor; glioblastoma multiforme; GBM; brain tumor; neuroendocrine tumor
MeSH Terms: conditions — Neoplasms; Glioblastoma; Brain Neoplasms; Neuroendocrine Tumors | interventions — dactolisib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BEZ235 and Everolimus (Experimental)
  Interventions: Drug: BEZ235; Drug: Everolimus

INTERVENTIONS:
Drug: BEZ235 — dose escalation 400mg- 1000mg per day
Drug: Everolimus — dose escalation 2.5 to 5 mg per day
  Other Names: RAD001

SUMMARY:
The purpose of this clinical trial is to determine the effects good or bad of combining BEZ235 along with Everolimus to determine if it is a safe treatment for patients with advanced cancers of different types.

DETAILED DESCRIPTION:
BEZ235 is an agent that was developed to slow down or halt cell growth and proliferation. It works by inhibiting two pathways that are important for cell growth and replication, one is called mTOR and the other is called PI3K.

Everolimus is an agent that also targets mTOR thus also slows down cell growth and spread; in addition, it injures blood vessels that supply cancer cells with nutrition.

The rationale behind combining Everolimus with BEZ235 is to inhibit cell growth and halt cancer spread by greater degree than either drug alone.

BEZ235 is not approved by the FDA for use in humans outside the context of a clinical trial.

Everolimus is FDA approved for the treatment of renal cell carcinoma (kidney cancer), subependymal giant cell astrocytoma (SEGA) associated with tuberous sclerosis (TS), and Advanced Neuroendocrine Tumors of Pancreatic Origin (PNET).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid malignancies that are metastatic or unresectable, and for which standard/curative measures do not exist by RECIST 1.1 measureable lesion which is not declining
* Age ≥ 18 years old at the day of consenting to the study
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate bone marrow and organ function as defined by laboratory values

Exclusion Criteria:

* Previous treatment with PI3K inhibitors
* Concurrent malignancy or has a malignancy within 3 years of study enrollment, (with the exception of adequately treated basal or squamous cell carcinoma or cervical carcinoma in situ)
* Concurrently using other approved or investigational antineoplastic agent
* Currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, hormonal therapy, etc.)
* Poorly controlled diabetes mellitus (HbA1c > 8 %)
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Active cardiac disease
* Inadequately controlled hypertension (i.e, SBP >180 mmHg or DBP >100mmHg)
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BEZ235 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea grade ≥ 2, malabsorption syndrome, or small bowel resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-01; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: John Morris, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Wise-Draper TM, Moorthy G, Salkeni MA, Karim NA, Thomas HE, Mercer CA, Beg MS, O'Gara S, Olowokure O, Fathallah H, Kozma SC, Thomas G, Rixe O, Desai P, Morris JC. A Phase Ib Study of the Dual PI3K/mTOR Inhibitor Dactolisib (BEZ235) Combined with Everolimus in Patients with Advanced Solid Malignancies. Target Oncol. 2017 Jun;12(3):323-332. doi: 10.1007/s11523-017-0482-9. PMID 28357727